CLINICAL TRIAL: NCT06317584
Title: The Establishment of "Empowerment-based Complementary and Alternative Medicine (ECAM) " Educational Program to Improve Complementary and Alternative Medicine(CAM) Health Literacy in Patients With Diabetes: Dilemma Analysis, Integration Into Practice and Outcome Evaluation
Brief Title: Empowerment-based Complementary and Alternative Medicine (ECAM)
Acronym: CAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiao-Yun Chang, professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: NMRPF3M0042
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: Complementary and Alternative Medicine (CAM); Patient Education; Empowerment; Health Literacy; Application; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Empowerment

STUDY DESIGN:
Intervention Model Description: Randomized trail method
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The process of keeping the study group assignment hidden after the allocation to participant, care provider, investigator, outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empowerment Application for CAM Health Education. (Experimental): Using empowerment software applications for complementary and alternative therapy education, explaining the risk factors that need to be considered, and teaching the use of the assistive tool of the empowerment software application
  Interventions: Other: Experimental: Empowerment Application for CAM Health Education
- Written Paper for CAM Health Education. (Placebo Comparator): Using written paper for complementary and alternative therapy education, explaining the risk factors that need to be considered
  Interventions: Other: Written Paper for CAM Health Education

INTERVENTIONS:
Other: Experimental: Empowerment Application for CAM Health Education — Using empowerment software application for complementary and alternative therapy education, explaining the risk factors that need to be considered, and teaching the use of assistive tool of the empowerment software application
  Arms: Empowerment Application for CAM Health Education.
Other: Written Paper for CAM Health Education — Using written paper for complementary and alternative therapy education and explaining the risk factors that need to be considered
  Arms: Written Paper for CAM Health Education.

SUMMARY:
This phase study will use a randomized trial method to evaluate the performance of the ECAM educational app in the promotion of CAM health literacy and communication among patients with diabetes.

DETAILED DESCRIPTION:
The objectives of this phase study are to (1) implement the ECAM educational app to empower patients with diabetes in their management of diabetes alongside CAM use; (2) examine the impact of the ECAM educational app on patient empowerment, CAM health literacy, risk management of CAM use, CAM communication and diabetes quality of life in patients with diabetes; and (3) collect feedback from both patients and nurses on how to improve the ECAM educational app for dissemination and implementation.

ELIGIBILITY:
Inclusion Criteria:

* People over the age of 20
* diagnosis of diabetes at least 12 months before the interview; and
* The use of CAM at least 3 months
* Sufficient mental ability to understand the informed consent form and sign it.

Exclusion Criteria:

* Participants will be excluded by an assistant researcher if they serious physical condition and hard of hearing and seeing.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Understanding the benefits-risks of complementary therapies (CTs) use scale Alternative Medicine (CAM) use questionnaire | Pre-test (baseline), 2, 3 months after intervention
  Measure patients' understanding of benefit-risk management on CAM use，The lower the score, the poorer the understanding.
Quality of life questionnaire | Pre-test (baseline), 2, 3 months after intervention
  assess patients' satisfaction with various aspects of life while managing diabetes.
Diabetes Empowerment scale | Pre-test (baseline), 2, 3 months after intervention
  Measure patients' understanding of benefit-risk management on CAM use, the minimum and maximum values，and higher scores .The minimum is 10，maximum values is 40，The lower the score, the poorer the understanding.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hsiao Yun, PhD, Study Chair — Chang Gung University of Science and Technology
Locations (1):
- CHENG GUNG MEMORIAL HOSPITAL, Linkou, Taoyuan, Guishan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.